CLINICAL TRIAL: NCT06915064
Title: Effect of Photobiomodulation in Patients With Temporomandibular Dysfunction Refractory to Botulinum Toxin Treatment: A Non-controlled Multicentric Pilot Study
Brief Title: Effect of Photobiomodulation in Patients With Temporomandibular Dysfunction Refractory to Botulinum Toxin Treatment.
Status: Completed | Type: Observational
Sponsor: University of Coimbra (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Principal Investigator, Bruno Macedo de Sousa, Professor, University of Coimbra
Other Study IDs: USUCLLT2025
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Temporomandibular disorders; low- level laser- photobiomodulation therapy; TMD; myofascial TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- LLLT-PBMT: Three patients (30%) received treatment on the left side and seven (70%) on the right side. The treatment was carried out using the EPIC X laser (BIOLASE®), which uses a solid-state diode as a semiconductor source of invisible infrared radiation.
  Interventions: Device: Low- level laser- photobiomodulation therapy

INTERVENTIONS:
Device: Low- level laser- photobiomodulation therapy — Three patients (30%) received treatment on the left side and seven (70%) on the right side. The treatment was carried out using the EPIC X laser (BIOLASE®), which uses a solid-state diode as a semiconductor source of invisible infrared radiation. The therapy was applied to the masticatory muscles (temporal, masseter, internal pterygoid), to trigger points discovered on palpation and to the intra-articular area of the TMJ (posterior portion through the external ear, superior portion and anterior portion). All patients included in the study underwent four sessions of PBMT-LLL for four consecutive weeks. T

SUMMARY:
The objective of this preliminary research was to identify the effect of low-level laser photobiomodulation therapy (LLLT-PBMT) in patients with myofascial temporomandibular disorders (TMDs), refractory to botulinum toxin (BTX) treatment.

Specifically, the hypothesis of LLLT-PBMT as a safe, low-cost, painless, and minimally invasive alternative therapy was proposed to improve complete muscle recovery and significantly reduce muscle paralysis in patients with masticatory muscle disorders previously treated with BTX. Additionally, different treatment alternatives were investigated, and a protocol was suggested for the application of LLLT-PBMT in myofascial TMDs and the pain associated with masticatory muscles, also analyzing its complications and negative effects

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with TMDs. Presence of unilateral or bilateral painful symptoms. Associated conditions: Bruxism, hypertrophy of the masticatory muscles, headaches
* Previous treatment with BTX:

Minimum of 3 doses (100 IU) Applied in masticatory muscles and intracapsular area No favorable results obtained

Exclusion Criteria:

* Patients without prior treatment of this type.
* Patients receiving treatment in the Pain Unit.
* Patients undergoing invasive treatments: Open surgery in the cervicofacial region or TMJ arthrocentesis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten female patients were included who attended the Department of Maxillofacial Surgery at the University Hospital Complex of Salamanca.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Severity and frequency of the symptoms | Baseline and four weeks after the treatment
  To evaluate both the severity and the frequency of the symptoms associated with TMJ disorders, the anamnestic index of Fonseca was used, considered a valid tool for diagnostic confirmation.
Pain Intensity | Baseline and four weeks after the treatment
  For the evaluation of pain, the visual analog scale (VAS) was used, which provides a subjective evaluation of pain, with a scale of values from 0 to 10 representing the intensity of pain in an ascending manner.
Pressure pain threshold | Baseline and four weeks after the treatment
  Pressure pain (PP) was measured using a pressure algometer (Wagner FPI 10®) that shows its strength during manual therapy on pressure points (tip of the algometer perpendicular to the muscle, maintaining the pressure which is progressively increased up to 1 kg/sec).

SECONDARY OUTCOMES:
Maximum mouth opening | Baseline and four weeks after the treatment
  To measure the maximum mouth opening (MMO), a digital gauge (Ubermann®) was used, taking two measurements, and the average was used for statistical analysis.
Depression and anxiety | Baseline and four weeks after the treatment
  The Depression Anxiety Stress Scales-21 (DASS-21) questionnaire was used to assess affective states through the 21 questions that make up the tool. Scores are reported as a total score (ranging from 0 to 63) and individual scores for three subscales (ranging from 0 to 21). Additionally, percentiles are calculated based on community samples. Each subscale score is classified into five severity levels: normal, mild, moderate, severe, and extremely severe.
Satisfaction with the treatment | Four weeks after the treatment
  The degree of satisfaction with the treatment received was evaluated in the patients. For this purpose, the Likert scale was used, a validated scale consisting of 5 items that evaluates attitudes, perceptions or levels of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Nanci Lopez-Valverde, PhD, Principal Investigator — University of Salamanca
Locations (1):
- Department of Maxillofacial Surgery at the University Hospital Complex of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No